CLINICAL TRIAL: NCT01637376
Title: Photodynamic Therapy (PDT) With Temoporfin for Non-Resectable Non-Small-Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants were enrolled
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 134367
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Carcinoma, Non-Small-Cell-Lung
Keywords: Lung neoplasms; Non Small cell lung carcinoma; Non small cell lung cancer; Large cell carcinoma; squamous cell carcinoma; adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Carcinoma, Large Cell; Carcinoma, Squamous Cell; Adenocarcinoma | interventions — temoporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Temoporfin — A single dose of 0.04 mg per kilogram of body weight of Temoporfin will be administered by slow intravenous injection into a deep vein (such as the antecubital vein) in not less than 6 minutes and will not be flushed with sodium chloride or any other aqueous solution.
  Other Names: Foscan

SUMMARY:
The purpose of this study is to evaluate the safety of I-PDT with Temoporfin for patients with Non-Resectable Non-Small-Cell Lung Cancer (NR-NSCLC). Several clinical studies suggested that photodynamic therapy (PDT) may be an effective treatment for patients with NR-NSCLC. PDT is a therapy where an external light source, such as laser, is used to activate a light-sensitive medicine to produce byproducts that can destroy cancer cells. In this study the investigators will use an experimental light sensitive medicine, Temoporfin, to perform interstitial PDT (I-PDT). In I-PDT, laser fibers are inserted into the tumor to activate the light-sensitive medicine.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age and older, male or female, of all races and ethnicities.
* Histologically confirmed non-small-cell lung cancer (NSCLC).
* Not a candidate for curative surgery.
* Not a candidate for curative concurrent chemoradiation therapy.
* Not a candidate or does not wish to receive curative radiation therapy.
* Not a candidate or does not wish to receive radiofrequency or microwave thermal ablation.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status < 2.
* The tumor is observable in CT with contrast.
* The tumor is accessible for unrestricted illumination of interstitial photodynamic therapy (I-PDT).
* Deemed likely to survive for at least 3 months.
* Patient is able and willing to provide written informed consent to participate in the study.
* If the subject is a female of childbearing potential, the subject is willing to take a pregnancy test and practice strict birth control (estrogen-containing oral contraceptives or an intrauterine device) throughout the study and for 3 months after Temoporfin administration. Women who have had a hysterectomy are exempt from these requirements.
* Subject is willing to remain in a controlled light exposure environment for a time period of at least 15 days.
* History of laboratory tests that meet the following criteria
* Hematocrit >= 33%, hemoglobin >= 11 g/dl

  * Platelet count > 70,000 per microliter
  * White blood count > 3,000 per microliter or ANC > 1500 per microliter
  * Creatinine: 0.8 to 1.4 mg/dL
  * Serum chloride: 101 to 111 mmol/L
  * Serum potassium: 3.7 to 5.2 mEq/L
  * Serum sodium: 136 to 144 mEq/L
  * Liver function test: albumin, bilirubin (direct/conjugated), ALT (alanine transaminase), AST (aspartate transaminade), GGT (gamma glutamyl transferase), ALP (alkaline phosphatase) within normal limits
  * BUN: 7 to 20 mg/dL

Exclusion Criteria:

* The tumor invades a major blood vessel.
* The tumor is not clearly shown on the CT image.
* The tumor size is larger than 5 cm when measured in a contrasted CT image according to RECIST v1.1.
* The location and extension of the tumor precludes an effective I-PDT.
* Patient with porphyria or other diseases exacerbated by light.
* Patient with hypersensitivity to Temoporfin or to any of its excipients.
* Patient with known allergies/hypersensitivity to porphyrins.
* Patient with a planned surgical procedure within the next 30 days.
* Patient with a coexisting ophthalmic disease likely to require slit-lamp examination within the next 30 days.
* Patient with existing therapy with a photosensitizing agent (Temoporfin, porphyrin or derivatives of porphyrin).
* Patient has received prior PDT to the proposed treatment site within the prior 3 months.
* Patient with known sensitivity to the CT contrast agent (Omnipaque), which would preclude the use of the CT contrast agent.
* History of poor renal function as demonstrated by serum creatinine and estimated glomerular filtration rate (eGFR) < 40 mL/min/1.73m2, which would preclude the using of the CT contrast agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of serious adverse events | 14 and 30 days post-therapy
  The specific aim of this pilot study is to evaluate the safety of CT-guided I-PDT with Temoporfin on patients with NR-NSCLC. Patient safety will be the primary endpoint. The safety of the intervention will be assessed at 14 and 30 days post-therapy. The primary outcome will be occurrence of Serious Adverse Events (SAE).

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Meek, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States